CLINICAL TRIAL: NCT04203342
Title: A Randomized,Double-blind,Vehicle-controlled, Parallel-design,Multiple-site Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Douglas Pharmaceuticals America Ltd) to Ketoconazole Cream 2% (Teva Pharmaceuticals USA Inc.) in the Treatment of Tinea Pedis.
Brief Title: A Therapeutic Equivalence Study of Ketoconazole Cream 2%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Douglas Pharmaceuticals America Ltd (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry); ACM Global Laboratories (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71864602
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2019-12

CONDITIONS: Tinea Pedis
Keywords: Tinea pedis; Ketoconazole
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be randomised, packaged and blinded by an independent packaging company.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketoconazole 2% cream (Douglas Pharmaceuticals America Ltd.) (Experimental): Subject will be randomized to either test product/active comparator/placebo comparator. Test product is Ketoconazole 2% cream manufactured by Douglas Pharmaceuticals America Ltd.
  Interventions: Drug: Experimental: Ketoconazole 2% Cream (Douglas Pharmaceuticals America Ltd.)
- Ketoconazole 2% cream (Teva Pharmaceuticals USA) (Active Comparator): Subject will be randomized to either test product/active comparator/placebo comparator. Active comparator is Ketaconazole 2% cream manufactured by Teva Pharmaceuticals USA.
  Interventions: Drug: Active comparator: Ketoconazole 2% Cream (Teva Pharmaceuticals USA)
- Placebo (Douglas Pharmaceuticals America Ltd.) (Placebo Comparator): Subject will be randomized to either test product/active comparator/placebo comparator. Placebo comparator is manufactured by Douglas Pharmaceuticals America Ltd.
  Interventions: Drug: Placebo comparator: Placebo (Douglas Pharmaceuticals America Ltd.)

INTERVENTIONS:
Drug: Experimental: Ketoconazole 2% Cream (Douglas Pharmaceuticals America Ltd.) — Topical treatment for tinea pedis. Subjects will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 +/- 4 days. Each subject is expected to receive 42 +/- 4 doses.
  Arms: Ketoconazole 2% cream (Douglas Pharmaceuticals America Ltd.)
Drug: Active comparator: Ketoconazole 2% Cream (Teva Pharmaceuticals USA) — Topical treatment for tinea pedis. Subjects will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 +/- 4 days. Each subject is expected to receive 42 +/- 4 doses.
  Arms: Ketoconazole 2% cream (Teva Pharmaceuticals USA)
Drug: Placebo comparator: Placebo (Douglas Pharmaceuticals America Ltd.) — Topical placebo to treatment for tinea pedis. Subjects will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 +/- 4 days. Each subject is expected to receive 42 +/- 4 doses.
  Arms: Placebo (Douglas Pharmaceuticals America Ltd.)

SUMMARY:
Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% in the Treatment of Tinea Pedis.

DETAILED DESCRIPTION:
A randomized, double-blind, vehicle-controlled, parallel-design, multiple-site study to evaluate the clinical (therapeutic) effet of a generic Ketoconazole Cream 2% (Douglas Pharmaceuticals America Ltd) compared with the reference standard Ketoconazole Cream 2% (Teva Pharmaceuticals USA Inc) in subjects with a microbiologically-confirmed, clinical diagnosis of tinea pedis. Approximately 675 subjects, male or female, 18 years or older, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-lactating female, 18 years of age or older
* Signed ICF meeting all criteria of current FDA regulations
* Female subject of childbearing potential must NOT be pregnant or lactating at Visit 1 (negative urine pregnancy test)
* Female subject of childbearing potential must agree to use of reliable method of contraception.
* Clinical diagnosis of tinea pedis predominantly in interdigital spaces
* Tinea pedis confirmed at baseline by positive KOH wet mount.
* Sum of clinical signs and symptoms score of target lesion at least 4; in addition target lesion must have a minimum score of at least 2 for erythema and a minimum score of at least 2 for either pruritis or scaling.

Exclusion Criteria:

* Females who are pregnant, lactating or planning to become pregnant during the study period.
* history of, or current psoriasis, lichen planus, or contact dermatitis involving the feet within the previous 12 months.
* history of dermatophyte infections with a lack of response to antifungal systemic or topical therapy (recurrent tinea pedis [i.e.more than 3 infections in the past 12 months] that were unresponsive to previous antifungal therapy).
* history of allergy, hypersensitivity, or intolerance to ketoconazole, other imidazoles, sulfites or any other component of the study product.
* confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.
* current uncontrolled diabetes.
* presence of any other infection of the foot or other disease process that, in the Investigator's opinion, may interfere with the evaluation of the subject's tinea pedis.
* known history of or current impaired wound healing, presence of peripheral vascular disease and/or trophic changes of the lower limbs to an extent that, in the opinion of the Investigator would make the subject unsuitable for the study or compromise subject's safety.
* Signficant history or current evidence of chronic infectious disease, system disorder, organ disorder, immunosuppression (due to disease or therapy, including history of organ transplant), or other medical condition that, in the opinion of the Investigator, would place the subject at undue risk by participating or compromise the integrity of the study data.
* Use of antipruritics, including antihistamines, within 72 hours prior to Visit 1.
* Use of topical corticosteroids, topical antibiotics or topical antifungal therapy (e.g. clotrimazole, econazole, fluconazole) within 2 weeks before Visit 1.
* Use of systemic (e.g. oral or injectable) antibiotics, systemic antifungal therapy, or systemic corticosteroids within 30 days before Visit 1. The use of intranasal, inhaled or ophthalmic corticosteroids for acute or chronic conditions (e.g. allergic conjunctivitis, asthma/COPD maintenance) is acceptable to the extent that, in the opinion of the Investigator, does not compromise safety of subject or integrity of the data.
* Use of oral terbinafine or itraconazole within 2 months before Visit 1.
* Use of immunosuppressive medication or radiation therapy within 3 months before Visit 1.
* Receipt of any drug as part of a research study within 30 days before Visit 1.
* Previous participation in this study.
* Employee of the Investigator or research centre or their immediate family members.
* Inability to understand the requirements of the study and the relative information or are unable or unwilling to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Therapeutic cure of tinea pedis | 2 weeks post-treatment (Day 56)
  The proportion of subjects in each treatment group with a Therapeutic Cure of tinea pedis at the test-of-cure visit conducted 2 weeks after the end of treatment (Day 56 +/- 4). Therapeutic cure is defined as having both a clinical and mycological cure of tinea pedis.

SECONDARY OUTCOMES:
Clinical cure of tinea pedis | 2 weeks post-treatment (Day 56)
  The proportion of subjects in each treatment group with a Clinical Cure at Day 56 +/- 4. Clinical Cure is defined as a total severity score of </= 2, with no individual severity score of >1. This is calculated using The Clinical Signs and Symptoms of Tinea Pedis rated by the Investigator using a standardized rating scale as follows:
  0=none (complete absence of any sign or symptom)
  1. Mild (slight)
  2. moderate (definitely present)
  3. Severe (Marked, intense).
  The following signs and symptoms will be rated:
  Signs = fissuring/cracking, erythema, maceration, and scaling Symptoms = pruritis and burning/stinging
Mycological cure of tinea pedis | 2 weeks post-treatment (Day 56)
  The proportion of subjects in each treatment group with a Mycological Cure of tinea pedis at Day 56 +/- 4. Mycological Cure is defined as having a negative KOH test AND a negative fungal culture.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Moore Clinical Research, Brandon, Florida
  - Moore Clinical Reseach, Tampa, Florida
- FXM Research International, Belize City, Belize